CLINICAL TRIAL: NCT04808219
Title: Causes of Traffic Collisions of Ambulance Cars at the Prague Emergency Medical Services
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: David Peran (Other Government)
Responsible Party: Sponsor-Investigator, David Peran, Head of the Education and Training Centre, Emergency Medical Service, Prague
Organization: Emergency Medical Service, Prague (Other Government)
Other Study IDs: ZZSHMP_001_2021
Record Dates: First submitted 2021-02-25; First posted 2021-03-22 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Traffic Collision; Transport Accident
Keywords: traffic collision; safety; ambulances; emergency medical services

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Driver: Ambulance driver who was involved in a traffic collision - video analysis of the collision records and in-depth interview aiming to find the cause of the collision.

SUMMARY:
The aim of the project is to increase the protection of patients, employees and the organization by means of data collection about traffic collisions of ambulance cars.

DETAILED DESCRIPTION:
Published research studies have shown not only that approximately half of Emergency Medical Services (EMS) providers show signs of severe fatigue before traffic collision, but also that drowsy or tired EMS providers are significantly more often injured at work. Among the circumstances and factors contributing to the collisions, including environmental, road or equipment factors, the real causes of the collisions remain unclear, but might be investigated through interviews with participating drivers. The aim is to increase the protection of patients, employees and the organization by collect data in both qualitative and quantitative ways and to identify factors and measurable variables that might lead to strengthen healthy driving habits under the blue lights. The factors associated with ambulance accidents are not similar to those of the general driving population. The in-depth analysis of the whole problem aims not only to clarify the causes of collisions, but especially to create prevention steps so that such situations occur as little as possible.

The methodology will use the so-called mixed design - a combination of in-depth interviews with participating members of collisions (employees, or patient / relative), data from the road-scans and qualitative data including measurable variables.

A video-analysis of the collision will be performed. All data will be recorded anonymously - each participant in the accident will receive a special number for coding, under which they will appear. Data will be presented both in descriptive statistics and after statistical analysis (chi square test for independence and Fischer's exact test at the level of significance = 0.05).

In terms of qualitative data, in-depth interviews and their coding will be performed using grounded theory (based on Strauss and Corbin methodology). The aim is to gain the same view of events and their actions as the members of the group.

The sample of participants depends on collision rate, which was 50 incidents in the year 2020 (expecting approx. 100 cases in 2 years).

ELIGIBILITY:
Inclusion Criteria:

* ambulance driver involved in a traffic collision of ambulance car
* consent to participate in the study
* video recording of the collision exists and can be used

Exclusion Criteria:

* disagreement with participating in the study
* video recording of the collision cannot be obtained

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ambulance drivers of the Prague Emergency Medical Services with traffic collision.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Severity of the collision | Through study completion, an average of 2 year or until collection of 100 observations in total.
  3 levels of collisions' severity were set: (1) minor collision outside the public road, (2) minor collision caused on a public road and (3) severe collision.
Time frame of the collision | Through study completion, an average of 2 year or until collection of 100 observations in total.
  The time frame of the collision - includes the interval in which the collision happened - (1) way to the patient, (2) transport of the patient, (3) handover of the patient, (4) way from the hospital to the base, (5) out of duty.

CONTACTS AND LOCATIONS:
Overall Officials: David Peran, Dr., Study Chair — Prague Emergency Medical Services; Jaroslav Pekara, Ph.D., Study Director — Prague Emergency Medical Services
Locations (1):
- Prague Emergency Medical Services, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chiu PW, Lin CH, Wu CL, Fang PH, Lu CH, Hsu HC, Chi CH. Ambulance traffic accidents in Taiwan. J Formos Med Assoc. 2018 Apr;117(4):283-291. doi: 10.1016/j.jfma.2018.01.014. Epub 2018 Feb 7. PMID 29428195
- [Background] Tanaka K, De Lorenzo RA. Lights and Siren: A Risky Business? Ann Emerg Med. 2019 Jul;74(1):110-111. doi: 10.1016/j.annemergmed.2019.01.026. Epub 2019 Feb 21. No abstract available. PMID 30797574
- [Background] Wolfberg DM. Red Lights and Siren: High risk, high liability, little reward. JEMS. 2017 Feb;42(2):18-9. No abstract available. PMID 29215247
- [Background] Watanabe BL, Patterson GS, Kempema JM, Magallanes O, Brown LH. Is Use of Warning Lights and Sirens Associated With Increased Risk of Ambulance Crashes? A Contemporary Analysis Using National EMS Information System (NEMSIS) Data. Ann Emerg Med. 2019 Jul;74(1):101-109. doi: 10.1016/j.annemergmed.2018.09.032. Epub 2019 Jan 12. PMID 30648537
- [Background] Murray B, Kue R. The Use of Emergency Lights and Sirens by Ambulances and Their Effect on Patient Outcomes and Public Safety: A Comprehensive Review of the Literature. Prehosp Disaster Med. 2017 Apr;32(2):209-216. doi: 10.1017/S1049023X16001503. Epub 2017 Jan 30. PMID 28134063